CLINICAL TRIAL: NCT02934061
Title: A Phase III, Multicenter, Randomized Study to Assess the Efficacy and Safety of 0,5 mg Tizaspray® Administered Intranasally Versus Sirdalud® 2 mg Tablets, in Patients With Acute Low Back Pain
Brief Title: Study to Assess the Efficacy and Safety of Tizaspray® Versus Sirdalud®, in Patients With Acute Low Back Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MDM S.p.A. (Other)
Collaborators: Opera CRO, a TIGERMED Group Company (Other); Latis S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TZSA2
Record Dates: First submitted 2016-10-07; First posted 2016-10-14 (Estimated); Last update posted 2018-01-16 (Actual); Status verified 2017-03

CONDITIONS: Low Back Pain
Keywords: Acute low back pain
MeSH Terms: conditions — Low Back Pain | interventions — tizanidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tizaspray® (Experimental): Tizaspray® administered intranasally in patients with acute low back pain
  Interventions: Device: Tizaspray® administered intranasally
- Sirdalud® (Active Comparator): Sirdalud® 2 mg tablets administered in patients with acute low back pain
  Interventions: Drug: Sirdalud® 2 mg tablets administered

INTERVENTIONS:
Device: Tizaspray® administered intranasally — 0,5 mg Tizaspray® administered intranasally
  Other Names: Tizaspray®
  Arms: Tizaspray®
Drug: Sirdalud® 2 mg tablets administered — Sirdalud® 2 mg tablets administered in patients with acute low back pain
  Other Names: Sirdalud®
  Arms: Sirdalud®

SUMMARY:
Open label, randomized, controlled, multicenter study with two parallel groups of patients

DETAILED DESCRIPTION:
This is a phase III, open label, randomized, controlled, multicenter study with two parallel groups of patients.

Tizaspray® 0.5 mg (a new pharmaceutical form, liquid nasal spray solution), is proposed in this trial as a ready to use treatment for short term therapy of painful muscle spasms as the acute low back pain.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 65 years old
2. Average low back pain intensity moderate to severe (≥ 60 mm in the VAS) at Visit 1
3. Positivity to Schober test (i.e. measure < 5 cm) at Visit 1
4. Acute low back pain started at least 24 hours prior to inclusion in the trial and more than 6 weeks after the last episode of acute low back pain
5. Negative pregnancy test for women of childbearing potential (to be performed at Visit 1) and use of an acceptable mean of contraception (condom or mechanical methods) in the previous 2 months and for whole duration of the study
6. Signed Informed Consent

Exclusion Criteria:

1. History of chronic low back pain
2. Current treatment with drugs having significant effects at the alpha2 receptors whether agonist (i.e., clonidine, methyldopa) or antagonist (i.e., phenothiazines, imipramine)
3. Current treatment with any other muscle relaxant or any drugs having muscle relaxant properties
4. Known allergies, hypersensitivity, or intolerance to tizanidine or paracetamol or any excipients used in their manufacture (included patients with known rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption)
5. Signs of nasal congestion, nasal polyps, mucosal lesions of the nostrils, postnasal drip of any etiology or any clinically significant nasal pathology that may affect the absorption of study medication or the assessment of safety
6. Evidence of clinically unstable disease, as determined by medical history, physical examination, that, in the Investigator's opinion, preclude entry into the study
7. Spinal surgery within 1 year of study entry
8. Evidence of clinical gastrointestinal malabsorption
9. Use of steroids within 3 months of study entry or any other long-term treatment with steroids
10. Use of NSAID's or other anti-inflammatory drugs 6 hours prior to study inclusion
11. Use of fluvoxamine or ciprofloxacin, or other inhibitors of CYP1A2 such as antiarrhythmics (amiodarone, mexiletine, propafenone), cimetidine, fluoroquinolones (enoxacin, pefloxacin, norfloxacin), rofecoxib, oral contraceptives, and ticlopidine
12. Use of hypnotics or other CNS depressants
13. Blood pressure <100/70 mmHg
14. History of lumbar spinal stenosis, fibromyalgia, or ankylosing spondylitis
15. Severe scoliosis
16. More severe pain in a region other than the lower back
17. Acute low back pain associated with chills or fever
18. Pregnancy, breast feeding
19. Treatment with another investigational agent within the last 30 days
20. Known or suspected history of alcohol or drug abuse based on medical history, physical examination, or the Investigator's clinical judgment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
"hand-to-floor" distance, Low Back Pain Intensity Scale (0 to 100 mm VAS), Schober test (positive/negative), Roland Disability Questionnaire (RDQ) | days: 1

SECONDARY OUTCOMES:
"hand-to-floor" distance, Low Back Pain Intensity Scale (0 to 100 mm VAS), Schober test (positive/negative), Roland Disability Questionnaire (RDQ) | days: 3
"hand-to-floor" distance, Low Back Pain Intensity Scale (0 to 100 mm VAS), Schober test (positive/negative), Roland Disability Questionnaire (RDQ) | days: 8

CONTACTS AND LOCATIONS:
Overall Officials: Doina Rosu, MD, Principal Investigator — SCM GADOS
Locations (1):
- Opera Contract Research Organization SRL, Timișoara, Timiș County, Romania

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Liddle SD, Baxter GD, Gracey JH. Chronic low back pain: patients' experiences, opinions and expectations for clinical management. Disabil Rehabil. 2007 Dec 30;29(24):1899-909. doi: 10.1080/09638280701189895. Epub 2007 May 4. PMID 17852259
- [Background] Frymoyer JW. Back pain and sciatica. N Engl J Med. 1988 Feb 4;318(5):291-300. doi: 10.1056/NEJM198802043180506. No abstract available. PMID 2961994
- [Background] van Tulder M, Becker A, Bekkering T, Breen A, del Real MT, Hutchinson A, Koes B, Laerum E, Malmivaara A; COST B13 Working Group on Guidelines for the Management of Acute Low Back Pain in Primary Care. Chapter 3. European guidelines for the management of acute nonspecific low back pain in primary care. Eur Spine J. 2006 Mar;15 Suppl 2(Suppl 2):S169-91. doi: 10.1007/s00586-006-1071-2. No abstract available. PMID 16550447
- [Background] Cabitza P, Randelli P. Efficacy and safety of eperisone in patients with low back pain: a double blind randomized study. Eur Rev Med Pharmacol Sci. 2008 Jul-Aug;12(4):229-35. PMID 18727454
- [Background] Gorska J. [Effects of back pain treatment with tizanidine]. Ortop Traumatol Rehabil. 2005 Jun 30;7(3):306-9. Polish. PMID 17611479
- [Background] Malanga GA, Dennis RL. Use of medications in the treatment of acute low back pain. Clin Occup Environ Med. 2006;5(3):643-53, vii. doi: 10.1016/j.coem.2006.03.002. PMID 16963380
- [Background] Bernstein E, Carey TS, Garrett JM. The use of muscle relaxant medications in acute low back pain. Spine (Phila Pa 1976). 2004 Jun 15;29(12):1346-51. doi: 10.1097/01.brs.0000128258.49781.74. PMID 15187636
- [Background] Von Korff M, Saunders K. The course of back pain in primary care. Spine (Phila Pa 1976). 1996 Dec 15;21(24):2833-7; discussion 2838-9. doi: 10.1097/00007632-199612150-00004. PMID 9112707
- [Background] Henschke N, Maher CG, Refshauge KM. A systematic review identifies five "red flags" to screen for vertebral fracture in patients with low back pain. J Clin Epidemiol. 2008 Feb;61(2):110-118. doi: 10.1016/j.jclinepi.2007.04.013. Epub 2007 Aug 27. PMID 18177783
- [Background] Vitale DC, Piazza C, Sinagra T, Urso V, Cardi F, Drago F, Salomone S. Pharmacokinetic characterization of tizanidine nasal spray, a novel intranasal delivery method for the treatment of skeletal muscle spasm. Clin Drug Investig. 2013 Dec;33(12):885-91. doi: 10.1007/s40261-013-0137-2. PMID 24085590
- [Background] Miettinen TJ, Kanto JH, Salonen MA, Scheinin M. The sedative and sympatholytic effects of oral tizanidine in healthy volunteers. Anesth Analg. 1996 Apr;82(4):817-20. doi: 10.1097/00000539-199604000-00024. PMID 8615503
- [Background] Berry H, Hutchinson DR. Tizanidine and ibuprofen in acute low-back pain: results of a double-blind multicentre study in general practice. J Int Med Res. 1988 Mar-Apr;16(2):83-91. doi: 10.1177/030006058801600202. PMID 2967781
- [Background] Fryda-Kaurimsky Z, Muller-Fassbender H. Tizanidine (DS 103-282) in the treatment of acute paravertebral muscle spasm: a controlled trial comparing tizanidine and diazepam. J Int Med Res. 1981;9(6):501-5. doi: 10.1177/030006058100900613. PMID 6459256
- [Background] Hennies OL. A new skeletal muscle relaxant (DS 103-282) compared to diazepam in the treatment of muscle spasm of local origin. J Int Med Res. 1981;9(1):62-8. doi: 10.1177/030006058100900111. PMID 6451461
- [Background] van Tulder MW, Touray T, Furlan AD, Solway S, Bouter LM. Muscle relaxants for non-specific low back pain. Cochrane Database Syst Rev. 2003;2003(2):CD004252. doi: 10.1002/14651858.CD004252. PMID 12804507